CLINICAL TRIAL: NCT07082023
Title: Comparison of V-NOTES (Vaginal Natural Orifice Transluminal Endoscopic Surgery) Mesh-Free Sacrocolpopexy and Laparoscopic Mesh-Free Sacrocolpopexy
Brief Title: Comparison of V-NOTES and Laparoscopic Mesh-Free Sacrocolpopexy Techniques
Acronym: vnotes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, md, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gopvnotessacrocolpopexy
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: Sacrocolpopexy; vNOTES
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, randomized, parallel-group clinical trial comparing two minimally invasive surgical techniques for pelvic organ prolapse repair: V-NOTES sacrocolpopexy and laparoscopic sacrocolpopexy, both performed without synthetic mesh. Participants will be randomly assigned (1:1) to either group. The study aims to evaluate outcomes using validated tools including POP-Q, PFDI-20, and PISQ-12 over a 6-month follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-NOTES Sacrocolpopexy (Experimental): Patients undergoing mesh-free sacrocolpopexy via vaginal natural orifice transluminal endoscopic surgery (V-NOTES).
  Interventions: Procedure: V-NOTES Mesh-Free Sacrocolpopexy
- Laparoscopic Sacrocolpopexy (Active Comparator): Patients undergoing mesh-free sacrocolpopexy via conventional laparoscopy.
  Interventions: Procedure: Laparoscopic Mesh-Free Sacrocolpopexy

INTERVENTIONS:
Procedure: V-NOTES Mesh-Free Sacrocolpopexy — Mesh-free sacrocolpopexy performed via vaginal natural orifice transluminal endoscopic surgery (V-NOTES).
  Arms: V-NOTES Sacrocolpopexy
Procedure: Laparoscopic Mesh-Free Sacrocolpopexy — Mesh-free sacrocolpopexy performed via conventional laparoscopy.
  Arms: Laparoscopic Sacrocolpopexy

SUMMARY:
This study aims to compare the surgical outcomes, safety profiles, and patient satisfaction between two minimally invasive techniques for pelvic organ prolapse repair: Vaginal Natural Orifice Transluminal Endoscopic Surgery (V-NOTES) mesh-free sacrocolpopexy and laparoscopic mesh-free sacrocolpopexy. By evaluating perioperative data, complication rates, anatomical and functional outcomes, this trial seeks to determine whether the V-NOTES approach provides comparable or superior results to the traditional laparoscopic technique, without the use of synthetic mesh.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common condition among women, especially with increasing age and parity, often requiring surgical intervention. Sacrocolpopexy is considered the gold standard for apical prolapse repair due to its high anatomical success rate and long-term durability. Traditionally performed via open or laparoscopic approaches, sacrocolpopexy has evolved with minimally invasive techniques.

Recently, mesh-related complications have led to a growing interest in mesh-free alternatives. Simultaneously, natural orifice approaches such as Vaginal Natural Orifice Transluminal Endoscopic Surgery (V-NOTES) have gained popularity due to better cosmetic results, reduced postoperative pain, and faster recovery times.

This prospective, comparative study aims to evaluate and compare the clinical outcomes of mesh-free sacrocolpopexy performed via V-NOTES versus the laparoscopic approach. Parameters including operative time, intraoperative and postoperative complications, hospital stay, pain scores, anatomical success, and patient satisfaction will be analyzed. The goal is to assess whether V-NOTES can be a safe and effective alternative to laparoscopic mesh-free sacrocolpopexy in the surgical management of POP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to Gaziosmanpaşa Education and Research Hospital, Gynecology and Obstetrics Clinic, who underwent surgery due to symptomatic pelvic organ prolapse with apical and anterior POP Q stage 2 and above, Being over 18 years old Patients who underwent surgery by experienced surgeons

Exclusion Criteria:

* Having previously received KT and/or RT due to any malignancy Having previously undergone surgery due to proplasus Patients with severe cardiovascular or respiratory disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pelvic Organ Prolapse Quantification (POP-Q) stage from baseline to 6 months | Baseline and 6 months postoperative
  Anatomical success will be evaluated using the POP-Q system. A reduction of prolapse stage by at least one level or achieving stage 0-1 will be considered successful.
Change in PISQ-12 Score | Baseline and 6 months postoperative
  Sexual function will be evaluated with PISQ-12. An increase in score indicates improvement.
Change in Pelvic Floor Distress Inventory-20 (PFDI-20) Score | Baseline and 6 months postoperative
  Patient-reported symptoms related to pelvic floor distress will be evaluated using the PFDI-20. A decrease in score indicates improvement in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: süleyman salman, prof, Study Director — Gaziosmanpaşa Training and Research Hospital; havva betül bacak, md, Principal Investigator — Gaziosmanpaşa Training and Research Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No